CLINICAL TRIAL: NCT00858793
Title: High-dose Chemotherapy With Transplantation of Gene-modified Haematopoietic Stem Cells for HIV-positive Patients With Malignant Diseases Indicating an HSCT
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A leukaemia case was reported in patient treated with a similar vector. For safety risk we stopped recruitment
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARL-GT 2005
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: AIDS-related Lymphoma; HIV Infections
Keywords: AIDS; HIV; Lymphoma; Stem Cell Transplantation; gene-modified Stem Cells; treatment experienced
MeSH Terms: conditions — Lymphoma, AIDS-Related; HIV Infections; Acquired Immunodeficiency Syndrome; Lymphoma | interventions — Genes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Procedure: PBSC-M87o, Gene (M87o)-modified, CD34+ peripheral blood progenitor cells (PBSC)

INTERVENTIONS:
Procedure: PBSC-M87o, Gene (M87o)-modified, CD34+ peripheral blood progenitor cells (PBSC) — Patient stem cells will be mobilized with induction chemotherapy (R)-ICE and G-CSF. If sufficient cells can be mobilized, patients will be treated with high-dose chemotherapy and a transplant of autologous CD34+ cells transduced with an antiviral vector (M87o). If autologous CD34+ yield is insufficient, allogeneic gene-modified cells will be given, if a compatible donor is available. To minimize risk of transplant failure, a second unmodified CD34+ cell transplant will be given one week after the first transplant.

SUMMARY:
Patient stem cells will be mobilized with induction chemotherapy (R)-ICE and G-CSF. If sufficient cells can be mobilized, patients will be treated with high-dose chemotherapy and a transplant of autologous CD34+ cells transduced with an antiviral vector (M87o). If autologous CD34+ yield is insufficient, allogeneic gene-modified cells will be given, if a compatible donor is available. To minimize risk of transplant failure, a second unmodified CD34+ cell transplant will be given one week after the first transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of any ethnic group aged between 18 and 65 years
* HIV-positive patients with malignant diseases of the blood (NHL, Hodgkin disease, plasmocytoma, acute and chronic leukaemia) who failed to achieve complete remission (CR) after standard-dose first-line chemotherapy or had a chemosensitive relapse after an initial CR
* Patients must receive HAART

Exclusion Criteria:

* Any of the following conditions:

  * congestive heart failure (NYHA > II)
  * documented EBV, HBV or HCV infection (only for allogeneic PBSCT)
  * creatinine clearance < 60 ml/min
  * left ventricular ejection fraction < 40%
  * bilirubin > 2 mg/dl
* Severe opportunistic infection
* More than 10% of bone marrow involved with lymphoma
* Between 2 and 5 10^6 autologous CD34+ cells/kg BW obtained after leukapheresis and CD34 enrichment
* Women of child.bearing potential not under adequate contraceptive protection
* Women who are pregnant or breast feeding
* Known history of drug-, medication- or alcohol abuse within the last 12 months preceding the study
* Participation in another study with an investigational product within less than one month prior to this study
* Simultaneous participation in a study with an investigational drug
* Presence of any disease likely to require procedures altering the schedule of the protocol
* Patients with a history of seizures, central nervous system disorders or psychiatric disability thought to be clinically significant in the opinion of the investigator
* Patients with limited mental capacity to the extent that he/she cannot provide informed consent or information regarding adverse events of the study medication
* Patients with any clinically meaningful renal, hepatic, respiratory or cardiovascular disease
* Patients who have previously been admitted to this study
* Patients who will not accept transfusions of blood products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-11-28 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Adverse events, ECOG performance status and laboratory safety tests | five years after transplantation

SECONDARY OUTCOMES:
Remission status (CR or PR) | five years after transplantation
Any relapse of ARL | five years after transplantation
level and kinetics of engraftment and level of gene marking | five years after transplantation
Viral load | five years after transplantation
CD4 counts | five years after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kroeger, Principal Investigator — University Medical Center Hamburg-Eppendorf, Department for Stem Cell Transplantation
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Result] Yla-Herttuala S. Gene therapy moves forward in 2010. Mol Ther. 2011 Feb;19(2):219-20. doi: 10.1038/mt.2010.307. No abstract available. PMID 21289631
- See also: page 1435; abstract 109 — https://www.esgct.eu/home/Previous%20Congresses/2010_Milan/Milan_2010_abstracts.pdf